CLINICAL TRIAL: NCT00888316
Title: Iron Overload in Allogeneic Hematopoietic Cell Transplantation
Brief Title: Iron Overload in Patients Undergoing Donor Stem Cell Transplant
Status: Completed | Type: Observational
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2008NTLS103; 0807M41481 (Other: IRB, University of Minnesota); CICL670AUS28T (Other: Novartis Pharmaceuticals)
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Cancer; Hematopoietic Stem Cell Transplantation; Allogeneic Hematopoietic Cell Transplantation
Keywords: iron overload
MeSH Terms: conditions — Neoplasms; Iron Overload | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Without Iron Overload: Patients entering study without pre-HSCT iron-overload. Iron overload will be defined as liver ion concentration (LIC above normal (>1.8 mg/g) on R2 magnetic resonance imaging (MRI) of the liver.
  Interventions: Procedure: magnetic resonance imaging; Procedure: Serum ferritin
- With Iron-Overload: Patients entering study with pre-HSCT iron-overload. Iron overload will be defined as liver ion concentration (LIC above normal (>1.8 mg/g) on R2 magnetic resonance imaging (MRI) of the liver.
  Interventions: Procedure: magnetic resonance imaging; Procedure: Serum ferritin

INTERVENTIONS:
Procedure: magnetic resonance imaging — MRI of the liver will be performed within 30 days prior to HSCT (day 0) and can be done during receipt of conditioning regimen chemotherapy and/or radiation therapy. MRI will also be performed in selected patients at 1 year post-HSCT. This MRI will be done within ± 30 days of their 1-year post-transplant followup date.
  The R2 MRI is a specific MRI technique and cannot be used for the purpose of general diagnostic imaging. In our study, this modality is being used specifically for the estimation of LIC.
  Other Names: R2 MRI
Procedure: Serum ferritin — Blood samples will be taken pre-transplant, 3, 6, 9 and 12 months post-transplant

SUMMARY:
RATIONALE: Learning about the effect of excess iron in the liver of patients undergoing donor stem cell transplant may help doctors plan treatment.

PURPOSE: This study is investigating the effects of iron overload in patients undergoing donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the impact of pre-transplant iron overload (defined as liver iron concentration [LIC] above normal [> 1.8 mg/g] on an MRI of the liver measuring tissue proton transverse relaxation rates [R2 MRI]) on the probability of 1-year overall survival of patients undergoing allogeneic hematopoietic stem cell transplantation (HSCT).

Secondary

* Determine the impact of pre-transplant iron overload on the composite endpoint of non-relapse mortality and complications (e.g., serious infections, hepatic veno-occlusive disease, or organ failure) within 1 year after allogeneic HSCT.
* Determine the impact of pre-transplant iron overload on the 1-year cumulative incidence of acute or chronic graft-vs-host disease in patients with acute leukemia or myelodysplastic syndromes undergoing allogeneic HSCT.
* Determine the impact of pre-transplant iron overload on the 1-year probability of overall survival and non-relapse mortality in patients undergoing allogeneic HSCT.
* Determine the prevalence of pre-transplant iron overload in adult patients undergoing allogeneic HSCT.
* Determine the correlation between pre-transplant ferritin levels and LIC on R2 MRI.
* Compare the longitudinal measures of serum ferritin levels after allogeneic HSCT in patients with iron overload vs those without iron overload.
* Estimate the cumulative incidence of iron overload at 1 year after allogeneic HSCT.

OUTLINE: Patients undergo blood sample collection to measure serum ferritin levels at baseline (pre-transplant) and then at 3, 6, 9, and 12 months after transplant. Patients with serum ferritin > 500 ng/mL also undergo an R2 MRI at baseline (pre-transplant) and at 12 months after transplant to determine liver iron concentration. Patients with serum ferritin > 500 ng/mL at 12 months after transplant also undergo an R2 MRI.

ELIGIBILITY:
Inclusion Criteria:

* Planning to undergo allogeneic hematopoietic stem cell transplantation using either myeloablative or reduced-intensity conditioning

  * Any diagnosis allowed
* Not pregnant
* Weight ≤ 350 lbs
* Must be able to give written informed consent indicating the investigational nature of the study and its potential risks.

Exclusion Criteria:

* Claustrophobia
* Other contraindication for MRI (e.g., cardiac pacemaker, implanted cardiac defibrillator, aneurysm clips, carotid artery vascular clamp, neurostimulator, insulin or infusion pump, or implanted drug infusion device)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Allogeneic Hematopoietic Cell Transplantation
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2008-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 1 Year
  Number of patients alive at 1 year.

SECONDARY OUTCOMES:
Incidence of non-relapse mortality | Up to 1 Year
  Number of patients who died due to serious infections, hepatic venous occlusive disorder (VOD) or organ failure within one year of transplant.
Acute and chronic graft-vs-host disease | 1 Year Post Transplant
  Number of patients who had acute and chronic graft versus host disease through 1 year after transplant.
Overall survival and non-relapse mortality | 1 Year Post Transplant
  Number of patients who were alive and did not have any non-relapse mortality events at 1 year post transplant.
  Determine the impact of pre-transplant iron-overload on 1-year probability of overall survival and of non-relapse mortality in allogeneic HSCT recipients with acute leukemia and myelodysplastic syndrome.
Number of Patients with Iron Overload | Baseline
  Prevalence of iron overload in patients being considered for allogeneic HSCT
Ferritin levels and Liver Iron Concentration | Baseline, and 3, 6, 9, and 12 Months Post Transplant
  Correlation between pre-transplant and post-transplant ferritin levels and liver iron concentration on an MRI of the liver measuring tissue proton transverse relaxation rates (R2 MRI)
Longitudinal averages of serum ferritin levels | Post Transplant
  Compare the longitudinal measures of serum ferritin between the no iron-overload and iron-overload groups.
Incidence of iron overload | 1 Year Post Transplant
  Compare the longitudinal measures of serum ferritin between the no iron-overload and iron-overload groups.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Burns, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Children's Hospital - Fairview, Minneapolis, Minnesota, United States